CLINICAL TRIAL: NCT00078767
Title: Pharmacologic Treatment of PTSD in Sexually Abused Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Judith Cohen, Principle Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K02MH001938 (NIH); K02MH001938 (NIH)
Record Dates: First submitted 2004-03-05; First posted 2004-03-08 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Depression; Anxiety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TF-CBT + sertraline (Experimental): Trauma-Focused CBT provided individually to youth and parent for 12 sessions (90 minute sessions; 45 minutes for youth; 45 minutes for parent); plus Sertraline provided in dosage titrated as clinically indicated by child psychiatrist blind to treatment assignment, from 50mg/day to a maximum dosage of 150 mg/day
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy; Drug: Sertraline Pill
- TF-CBT +placebo (Active Comparator): Trauma-Focused CBT provided individually to youth and parent for 12 sessions (90 minute sessions; 45 minutes for youth; 45 minutes for parent); plus placebo identical to Sertraline, provided in pill form and titrated as clinically indicated by child psychiatrist blind to treatment assignment, from 1 to 3 pills/day (identical in appearance to 50 to 150mg/day of Sertraline)
  Interventions: Drug: Sertraline Pill; Drug: Placebo Oral Tablet

INTERVENTIONS:
Behavioral: Trauma-Focused Cognitive Behavioral Therapy — 12 weeks of Trauma-Focused CBT (TF-CBT)for youth and parent
  Arms: TF-CBT + sertraline
Drug: Sertraline Pill — 12 weeks of Sertraline pill, flexible dosage of 50-150 mg/day, to be administered while receiving TF-CBT
Drug: Placebo Oral Tablet — 12 weeks of Placebo pill, flexible dosage, of 50-150 mg/day, to be administered while receiving TF-CBT
  Arms: TF-CBT +placebo

SUMMARY:
This study will evaluate the benefit of adding sertraline (Zoloft®) to Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) for sexually abused children who have Posttraumatic Stress Disorder (PTSD).

DETAILED DESCRIPTION:
Adult research has demonstrated the efficacy of selective serotonin reuptake inhibitors (SSRIs) in decreasing Posttraumatic Stress Disorder (PTSD) symptoms; to date the SSRIs are the only medication class with demonstrated efficacy in treating all three PTSD symptom clusters (reexperiencing, avoidance, and hyperarousal). No studies have evaluated the impact of SSRIs on PTSD symptoms in children or adolescents. Trauma-focused CBT has been shown in several studies to be efficacious in decreasing PTSD symptoms in sexually abused children and adolescents. Many children and youth with PTSD are currently prescribed SSRIs and other medications. This study will evaluate whether adding the SSRI sertraline provides additional benefits over TF-CBT treatment for sexually abused children and adolescents with PTSD. If adequate numbers of children with comorbid PTSD and depressive and/or anxiety disorders are included, it may also be possible to evaluate whether any benefit of adding sertraline is restricted to those children with comorbid disorders.

ELIGIBILITY:
Inclusion:

1. Ages 10-17 years, inclusive
2. Confirmed sexual abuse
3. At least 5 PTSD symptoms on KSADS-PL, with at least one symptom in each of 3 symptom clusters (reexperiencing, avoidance, arousal)
4. Parent/primary caregiver available to participate in treatment
5. Assent with parental consent to participate

Exclusion:

1. Non-English speaking
2. schizophrenia or other severe psychotic disorder
3. MR (IQ<60) or PDD preventing CBT treatment
4. taking current psychotropic medication
5. documented substance dependence (substance abuse allowed)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2001-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Cohen, M.D., Principal Investigator — Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Locations (1):
- Allegheny General Hospital Center for Traumatic Stress in Children and Adolescents, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Cohen JA, Mannarino AP, Perel JM, Staron V. A pilot randomized controlled trial of combined trauma-focused CBT and sertraline for childhood PTSD symptoms. J Am Acad Child Adolesc Psychiatry. 2007 Jul;46(7):811-9. doi: 10.1097/chi.0b013e3180547105. PMID 17581445
- See also: National Child Traumatic Stress Network — http://www.nctsnet.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TF-CBT + Sertraline | TF-CBT +Placebo
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TF-CBT + Sertraline | TF-CBT +Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 14 [10 to 17] | 14 [10 to 17] | 14 [10 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 6 | 12
  African American | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Kiddie-Sads-Present and Lifetime (KSADS-PL) Scale for PTSD
Description: Change in PTSD parameters as determined by changes in score. At enrollment, participants either did or did not have a PTSD diagnosis. The three categories displayed show participants who had the PTSD diagnosis at the time of enrollment but did have evidence of PTSD at the end of their participation, participants who had PTSD at enrollment and who continued to exhibit PTSD at the end of their participation, and those who did not have a PTSD diagnosis at the start of the trial. There are numerous criteria used to determine a PTSD diagnosis; they are not individually listed. The diagnosis was sufficient for the purposes of the study.
Time Frame: Up to 39 months
Measure: Count of Participants; unit: Participants
Arm/Group | TF-CBT + Sertraline | TF-CBT +Placebo
Number analyzed (Participants) | 11 | 11
Participants
  PTSD diagnosis at enrollment but no PTSD at end | 8 | 6
  PTSD at enrollment and PTSD at end | 1 | 5
  No PTSD diagnosis at enrollment and no PTSD at end | 2 | 0

2. Secondary Outcome: Mood and Feelings Questionnaire (MFQ) for Depressive Symptoms
Description: Change in depressive symptoms as determined by change in score
Time Frame: Up to 39 months
Population: There were two categories of depression: participants that had clinical signs of depression at the time of enrollment, and participants that did not have clinical signs of depression. Participants in the "clinical symptom present at enrollment" category were tested to see if their status changed during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | TF-CBT + Sertraline | TF-CBT +Placebo
Number analyzed (Participants) | 11 | 11
Participants
  Clinical symptoms CS at enrollment to no CS at end | 8 | 5
  No clinical symptoms at enrollment; no CS at end | 3 | 6

3. Secondary Outcome: Anxiety Symptoms
Description: Change in SCARED scores between treatment groups.There were two categories of depression: participants that had clinical signs of depression at the time of enrollment, and participants that did not have clinical signs of depression. Participants in the "clinical symptom present at enrollment" category were tested to see if their status changed during the trial.
Time Frame: Up to 39 months
Population: There were two categories of anxiety symptoms: participants that had clinical signs of anxiety at the time of enrollment as evidenced by their SCARED scores, and participants that did not have clinical signs of depression. Participants with clinical symptoms category were tested to see if their status changed during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | TF-CBT + Sertraline | TF-CBT +Placebo
Number analyzed (Participants) | 11 | 11
Participants
  Cinical at start to nonclinical at end of trial | 8 | 5
  Nonclinical at start of trial | 2 | 2
  Clinical at start and remained clinical | 1 | 4

4. Secondary Outcome: Global Impairment
Description: Change in Children's Global Assessment Scale (CGAS) between the two groups
Time Frame: Up to 39 months
Population: There were two categories of depression: participants that had clinical signs of impairment at the time of enrollment as evidenced by their CGAS scores, and participants that did not have clinical signs of depression. Participants clinical symptoms were tested to see if their status changed during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | TF-CBT + Sertraline | TF-CBT +Placebo
Number analyzed (Participants) | 11 | 11
Participants
  Clearly impaired to not clearly impaired | 9 | 6
  Remained clearly impaired | 2 | 5

5. Secondary Outcome: Incidence of Suicidality
Description: Change in degree of suicidal ideation during study
Time Frame: Up to 39 months
Measure: Count of Participants; unit: Participants
Arm/Group | TF-CBT + Sertraline | TF-CBT +Placebo
Number analyzed (Participants) | 11 | 11
Participants
  Suicigal ideation at start of trial | 4 | 1
  Suicidal ideation at end of trial | 0 | 0
  No suicidal ideation at start or end of trial | 7 | 10

ADVERSE EVENTS:
Time Frame: 39 months
Arm/Group | TF-CBT + Sertraline | TF-CBT +Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes